CLINICAL TRIAL: NCT06353620
Title: Structural-functional Connectome With High-density Electroencephalography in Drug-resistant Epilepsies and Rare Neurodevelopmental Syndromes With Epilepsy
Brief Title: Structural-functional Connectome in Drug-resistant Epilepsies and Neurodevelopmental Syndromes With Epilepsy
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 1018
Record Dates: First submitted 2024-03-20; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy; Angelman Syndrome; Dup15q Syndrome
MeSH Terms: conditions — Epilepsy; Angelman Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Epilepsy: EEG resting state recording, neuropsychological evaluation
  Interventions: Diagnostic Test: High Density EEG recording; Diagnostic Test: Rey Complex Figure Test
- Angelman Syndrome: EEG resting state recording, neuropsychological evaluation
  Interventions: Diagnostic Test: High Density EEG recording; Diagnostic Test: Rey Complex Figure Test
- Dup15q Syndrome: EEG resting state recording, neuropsychological evaluation
  Interventions: Diagnostic Test: High Density EEG recording
- Control Group: EEG resting staterecording
  Interventions: Diagnostic Test: High Density EEG recording

INTERVENTIONS:
Diagnostic Test: High Density EEG recording — Recording of resting state high density EEG (128 channels)
Diagnostic Test: Rey Complex Figure Test — Memeory functioning evaluation
  Groups: Angelman Syndrome; Epilepsy

SUMMARY:
Recent studies have shown that the aperiodic part of the signal (neuronal avalanches) of electroencephalography (EEG) contains important information about the dynamics of neuronal networks. Indeed, this has helped to identify functionally altered areas in patients with temporal epilepsy by simply using the resting EEG signal. Furthermore, it has been seen that the propagation of neuronal avalanches (VNs) correlates with the morphological organization of the cerebral cortex. Therefore, NAs represent a measure with direct utility for studying functional reorganization pre and post drug/surgical treatment. In addition, the aperiodic portion of the signal may represent a noninvasive measure of the excitation/inhibition relationship, which is known of being altered both in epilepsy and in some rare neurodevelopmental syndromes (example: Angelman and Dup15q)

DETAILED DESCRIPTION:
Electroencephalography is the tool of choice for the diagnosis of epilepsy. Its use is increasing in the clinic, especially in its high-density form (HD-EEG), because it can be used as a neuroimaging tool, supporting the process of identifying the epileptogenic network (NE) and monitoring the evolution of brain connectivity over time in relation to the epileptic process.In particular, the reorganization of the functional connectome following pharmacological and/or surgical treatment of epilepsy is an aspect that is still little studied, but it could represent a useful prognostic factor that can improve the clinical management of the affected person. In addition, high-density EEG can be applied for the purpose of characterizing functional brain connectivity in some rare neurodevelopmental diseases, particularly Angelman syndrome and Dup15q syndrome, pathological increasingly being studied as a model of neurodevelopmental, cognitive and behavioral alterations in addition to epilepsy. Relatively to recent developments of potentially "disease modifying" therapies for these pathologies, there is indeed a need for markers of brain functioning useful to objectively monitor clinical development.

The present study involves the systematization of data from noninvasive clinical-instrumental assessments such as EEG and structural MRI, acquired during the diagnosis process in drug-resistant epilepsies and rare neurodevelopmental syndromes associated with epilepsy, in order to analyze the relationship between functional-structural organization of the brain system and clinical aspects, including cognitive and behavioral functioning. In the context of epilepsy, a data collection will be carried out to which recent analytical approaches related to the study of the functional connectome will be applied, with the aim of characterizing the reorganization of brain networks over time, hypothesizing a process of progressive "normalization" of these in subjects who present, after the course of treatment (pharmacological and/or surgical), total freedom or a significant reduction of seizures. In parallel, the relationship between the organization of functional networks and cognitive/behavioral functioning pre- and post-treatment will be analyzed, in order to obtain a dynamic and longitudinal view of the patients' clinical evolution. With this in mind, it is important to understand that functional activity is intrinsically linked to brain structures, and in fact the project takes into account the anatomo-functional relationship of the connectome. This relationship is crucial in rare neurodevelopmental syndromes, such as Angelman syndrome and Dup15q, where the use of the structural-functional connectome is a relevant novel element for the purpose of characterizing a highly complex picture that disrupts the global development of the affected child/person. Indeed, the relationship between changes in functional relationships between brain areas and underlying physical connections, as well as the relationship between these and neurodevelopment, are still poorly understood. The second goal of the project is therefore to generalize the use of these patient-friendly methods, starting with data collected with noninvasive instrumentation, in order to improve the characterization of the neurocognitive profile, as well as a useful tool to identify syndrome-specific biomarkers to be used in monitoring clinical development.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of focal or generalized epilepsy, Angelman syndrome, or Dup15q, confirmed by specialist evaluation;
* at least one MRI scan of the brain that includes 3D T1 sequences;
* at least one 128-channel HD-EEG recording; and
* age between 6 and 75 years at the time of the evaluation of the present study;
* ability to take part in a neuropsychological evaluation.

Exclusion Criteria:

* vascular causes or non-low-grade tumors as causes of epilepsy;
* age different from the range 6-75 years;
* neuroradiological examination not complete (absence T1 3D);
* absence of HD-EEG 128-channel recording
* inability to take part in a neuropsychological evaluation.

Ages: 6 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of focal or generalized epilepsy, Angelman syndrome, or Dup15q
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Differences in the network coherence values in theta and alpha band after treatment | 2 years
  The outcome 1 one will be finalized to measures the changes of the coherence values before and after the treatment. Coherence is a measure defining the strength of functional connectivity between two brain regions. The pre- and post-treatment changes will be investigated specifically in the theta and alpha EEG frequency band, since these two bands are the most affected in epilepsy condition.
Stability of the alpha frequency band in the EEG activity | 2 years
  The detrend fluctuation analysis (DFA) in the alpha band of the EEG power spectrum provides information on excitatory and inihibitory balance of neural activity. For the outcome 2, the exponent of the DFA in the alpha band will be compared between patients with rare neurodevelopmental disorders (Angelman and Dup15q) vs. the healthy control group.
Correlation of neural excitation and memory performance | 2 years
  Correlation between the aperiodic component of the EEG power specturum with the memory functioning obtained with the Rey Complex Figure Test, pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco Duma, Principal Investigator — IRCCS E. Medea
Locations (1):
- IRCCS E.Medea, Conegliano, Treviso, Italy

IPD SHARING:
Plan to Share IPD: No